Study Protocol: Impact of perioperative body temperature on postoperative complications and pain in Video-assisted thoracoscopic surgery patients utilizing continuous temperature monitoring

Version 1.0

**Document Date: Jun 20th 2025** 

### 1. Study Title

Impact of perioperative body temperature on postoperative complications and pain in Video-assisted thoracoscopic surgery patients utilizing a continuous temperature monitoring System: A Prospective Cohort Study

## 2. Study Summary

# 2.1 Primary Objective

To investigate the impact of intraoperative hypothermia on postoperative complications (e.g., infections, cardiopulmonary events, prolonged hospitalization) in Video-assisted thoracoscopic surgery (VATS) patients.

## 2.2 Secondary Objective

To analyze the relationship between intraoperative hypothermia and the incidence of moderate-to-severe postoperative pain.

# 3. Study Design

Type: Prospective cohort study

Exposure Group: Intraoperative hypothermia (body temperature <36.0°C for ≥30 min at any time during surgery)

Non-Exposure Group: Body temperature consistently ≥36.0°C

Sample Size: 144 participants (72 per group; accounting for 10% dropout)

# 4. Participants

### 4.1 Inclusion Criteria:

- Age ≥18 years
- American society of anesthesiology (ASA) class I-III
- BMI 18.5-30 kg/m<sup>2</sup>
- Scheduled for VATS lung/mediastinal tumor resection (duration ≥1 hour)
- Receiving general anesthesia + regional block (TPVB + SAPB)
- Written informed consent

#### 4.2 Exclusion Criteria:

- Preoperative fever (>37.5°C) or hypothermia (<36.0°C); ASA ≥IV
- Chronic opioid use (>3 months), chronic pain, or immunosuppression
- Emergency surgery or conversion to thoracotomy
- Planned surgery <1 hour or requiring cardiopulmonary bypass
- Failed regional block (sensory block not covering T2–T8 at 4h postoperation)
- Thyroid dysfunction or neurological disorders affecting pain assessment

#### 5. Interventions/Monitoring

Temperature Monitoring: Wireless axillary sensor (non-surgical side), recorded every 5 minutes.

Hypothermia Management: Active warming (forced-air warmer + IV fluid warming) if temperature <36.0°C for ≥30 min.

Regional Block: Ultrasound-guided TPVB + SAPB.

Postoperative Analgesia: PCA with oxycodone (no basal infusion; 5mg bolus, 10-min lockout) + IV flurbiprofen (if no contraindication).

#### 6. Outcome Measures

- Primary outcome: Incidence of Clavien-Dindo grade ≥ II complications (Daily clinical review until discharge)
- Secondary outcome: Moderate-severe pain (NRS ≥4) at 24h/48h/72h/post-discharge; length of stay; ICU admission rate; 30-day readmission rate.

# 7. Follow-Up Schedule

| Timepoint | Assessments | Endpoint Focus |
|---|---|---|
| Postop 6h | NRS pain score; Rescue | Acute pain incidenc |
| | analgesia | |
| Postop 24h/48h/72h | NRS pain score; | Pain trajectory; Early |
| | Complications; | complications |
| | Drain/ambulation | |
| Discharge | Total LOS; Analgesia use | Hospitalization duration |
| Postop Day 7 | Wound healing; Unplanned | Wound complications |
| | visits | |
| Postop Day 30 | Complications; Chronic pain | 30-day morbidity; Persistent |
| | (NRS≥3) | pain |

# 8. Statistical Analysis

- Primary Analysis: Multivariable logistic regression (hypothermia  $\rightarrow$  complications), Kaplan-Meier for time-to-event.
- Secondary Analysis:
  - Logistic regression (hypothermia → pain), adjusted for regional block.
  - Interaction testing ("hypothermia × block efficacy").
  - Subgroup analysis by block success level.
- Software: R/Prism 8; Significance: p<0.05 (two-sided).

### 9. Ethics & Quality Control

- Ethics Approval: PKUPH IRB review prior to enrollment.
- Blinding: Outcome assessors masked to temperature group.
- Participant Protection: Voluntary withdrawal; anonymized data.

## 10. Timeline

- Preparation: Mar-May 2025 (IRB/registration/pilot)

- Enrollment: Jul 2025-Jun 2027

Analysis: Jul-Aug 2027Publication: Dec 2027